CLINICAL TRIAL: NCT02793947
Title: Efficacy of Peri-Incisional Multimodal Drug Injection Following Operative Management of Femur Fractures: A Randomized Controlled Trial
Brief Title: Efficacy of Peri-Incisional Multimodal Drug Injection Following Operative Management of Femur Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Michael C Willey, Clinical Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201501822
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative; Femur Fracture
Keywords: Peri-incisional injection; Multimodal analgesia; Femur fracture
MeSH Terms: conditions — Pain, Postoperative; Femoral Fractures | interventions — Ropivacaine; Epinephrine; Morphine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peri-incisional injection (Experimental): A 100 cc multimodal analgesic cocktail will be injected into the superficial and deep peri-incisional tissues after the completion of femur fracture fixation/instrumentation while the patient remains under general anesthesia and prior to wound closure. This cocktail includes 400 mg of 0.75% ropivacaine (53.33 mL), 0.6 mg of 1 mg/mL epinephrine (0.6 mL), 5 mg of 0.5 mg/mL morphine sulfate (10 mL), and 36.07 mL 0.9% sodium chloride solution. All infiltrations will be completed with a blunt trochar to minimize the risk of intravascular injection.
  Interventions: Drug: Ropivacaine; Drug: Epinephrine; Drug: Morphine; Drug: 0.9% sodium chloride solution
- Control (no injection) (No Intervention): Femur fracture fixation/instrumentation will be completed per the standard of care. No peri-incisional injection will be completed.

INTERVENTIONS:
Drug: Ropivacaine — 400 mg of 0.75% ropivacaine (53.33 mL) will be included in the multimodal analgesic cocktail that will be injected intra-operatively into the superficial and deep peri-incisional tissues after completion of femur fracture fixation/instrumentation.
  Other Names: Naropin
  Arms: Peri-incisional injection
Drug: Epinephrine — 0.6 mg of 1 mg/mL epinephrine (0.6 mL) will be included in the multimodal analgesic cocktail that will be injected intra-operatively into the superficial and deep peri-incisional tissues after completion of femur fracture fixation/instrumentation.
  Other Names: Adrenalin
  Arms: Peri-incisional injection
Drug: Morphine — 5 mg of 0.5 mg/mL morphine sulfate (10 mL) will be included in the multimodal analgesic cocktail that will be injected intra-operatively into the superficial and deep peri-incisional tissues after completion of femur fracture fixation/instrumentation.
  Other Names: Duramorph
  Arms: Peri-incisional injection
Drug: 0.9% sodium chloride solution — 36.07 mL 0.9% sodium chloride solution will be included in the multimodal analgesic cocktail that will be injected intra-operatively into the superficial and deep peri-incisional tissues after completion of femur fracture fixation/instrumentation.
  Other Names: 0.9% normal saline
  Arms: Peri-incisional injection

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a peri-incisional multimodal injection for post-operative pain control following operative management of femur fractures. Enrolled subjects will be prospectively randomized into either the peri-incisional injection or control cohorts. Patients will be treated with standard of care surgical techniques by the treating orthopaedic surgeon for the patient's specific fracture pattern. The patients randomized into the injection cohort will receive an intra-operative injection with 400 mg ropivacaine, 0.6 mg epinephrine, 5 mg and morphine into the local superficial and deep peri-incisional tissues while under general anesthesia. Visual analog pain scores will be collected every 4 hours after surgery for the first two post-operative days. Total narcotic consumption will also be recorded over eight hour intervals for the first two post-operative days. Medication related side effects will be monitored. The investigators hypothesize that the peri-incisional injection cohort will demonstrate an improved pain profile and utilize less parenteral narcotic analgesia in the early post-operative period.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy and safety of a peri-incisional multimodal injection for post-operative pain control following operative management of femur fractures. Patients will be identified by way of direct presentation to the orthopaedic trauma service with an acute femur fracture. If the patient meets the parameters for study enrollment (inclusion/exclusion criteria) the patient will be approached for introduction of the study by a member of the surgical team. If the patient is agreeable to study enrollment, he/she will have to complete the written informed consent process. This study protocol has received formal approval from the University of Iowa Institutional Review Board.

The study design is a prospective, randomized, double-blind comparative trial. Patients will be randomly assigned to the two treatment groups: peri-incisional multimodal injection and control (no injection). In order to create balanced cohorts with respect to intervention, randomization will be completed in a block format across six discrete surgical techniques: proximal femur open reduction and internal fixation (dynamic hip screw, trochanteric stabilizing plate), distal femur open reduction and internal fixation (lateral peri-articular locking plate), cephalomedullary fixation, other intramedullary fixation (antegrade or retrograde intramedullary device without fixed angle construct into the femoral head), percutaneous fixation, and arthroplasty (hemiarthroplasty or total hip arthroplasty). Randomization will be performed with use of Microsoft Excel (Microsoft, Redmond, Washington) to generate random numbers. The patients enrolled in the investigation as well as the nursing staff performing the post-operative assessments are blinded to treatment allocation.

Each patient will be treated with standard of care techniques chosen by the treating surgeon regardless of whether or not the patient decides to enroll in the study. Written informed consent will be obtained for the surgical procedure in addition to and independent from the study consent. All surgical procedures will be completed under general anesthesia. No spinal, regional, or preemptive anesthesia/analgesic regimen will be employed per study protocol. Surgical drain placement and pharmacologic venous thromboembolism prophylaxis will not be standardized. Post-operative pain management will continue per the institutional standard of care with a combination of intravenous and oral narcotic analgesia. The post-operative pain regimen will not be specified nor altered by the study protocol.

Patients randomized to the peri-incisional injection cohort will receive a single intra-operative injection while the subject is under general anesthesia following completion of fracture fixation/instrumentation. The local anesthetic cocktail includes 400 mg of 0.75% ropivacaine (53.33 mL), 0.6 mg of 1 mg/mL epinephrine (0.6 mL), 5 mg of 0.5 mg/mL morphine sulfate (10 mL), and 36.07 mL 0.9% sodium chloride solution. All pharmacologic agents in the anesthetic cocktail are FDA approved. For intra-articular proximal femur procedures the cocktail will be evenly distributed between the deep (synovium, capsule, periosteum, gluteus musculature) and superficial (fascia lata, vastus lateralis, subcutaneous plane) tissues prior to wound closure. The same pattern will be followed for extra-articular proximal femur procedures without direct injection of the synovium and capsule. The injection will be similarly distributed between the deep (synovium, capsule, periosteum) and superficial (quadriceps musculature, subcutaneous plane) tissues prior to wound closure for distal femur procedures. Injections for intramedullary nails will be placed around the nail entry site into bone and into the superficial tissues at both the entry site and cross lock locations. All infiltrations will be completed with a blunt trochar to minimize the risk of intravascular injection.

The primary outcome is visual analog pain scores over the first two post-operative days. Patients will be instructed to use a 10-cm visual analog scale to describe their current level of comfort with end points of zero corresponding to "no pain" and ten corresponding to "the most extreme possible pain." Pain assessments will be completed while patients are at rest at standardized intervals immediately prior to surgery, in the post-anesthesia care unit (captured as the mean of all individual data points), and every 4 hours following surgery for the first two post-operative days. Visual analog pain scores are collected and charted by nursing staff on the inpatient ward. All nursing staff will remain blinded to the treatment allocation. Physician staff that have knowledge of the intra-operative treatment and randomization are not involved in recording any outcome measures.

The secondary outcome measures are total narcotic consumption, wound complications, and drug-related side effects. Narcotic consumption will be recorded every eight hours for the first two post-operative days and transformed into narcotic equivalents. Every fifteen minutes in the post-anesthesia care unit and every four hours for the first two post-operative days nursing personnel will monitor the patients via direct observation and query for medication side effects related to ropivacaine toxicity including blurred vision, hearing problems, transient peripheral paralysis, dizziness, convulsion, uncontrolled muscle contraction, hypotension, bradycardia, and new onset arrhythmia. Anesthesiology staff will also perform two standardized post-operative assessments in the recovery room and on the first post-operative day to screen for adverse effects related to the injection.

An a priori power analysis was completed for sample size determination for the primary outcome measure. A preliminary retrospective analysis revealed a standard deviation of 2.5 on the visual analog pain scale twelve hours following surgery (unpublished data). Prior literature has suggested that a change of 1.0-1.3 points on the visual analog scale is clinically significant. Therefore, the investigators determined a total of 44 patients were required per study group in order to detect a 1.5 point difference on the visual analog scale with a power of 80% and a P-value of 0.05. The Student t test and the chi-squared test of association will be used to compare continuous and categorical variables between the two groups, respectively. Statistical significance is defined as p <0.05.

Patient confidentiality will be maintained at all times. Only approved research team personnel will review the medical records. Only the minimal data necessary to answer the research questions will be obtained. Collected electronic data will be stored on password protected servers. Written informed consent documents will be stored in a locked filing cabinet in the Department of Orthopaedics and Rehabilitation at the University of Iowa Hospitals and Clinics. Upon publication and completion of data analysis all information with patient identifiers will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sustained an acute femur fracture in any anatomic region (subcapital, basicervical, intertrochanteric, subtrochanteric, diaphyseal, distal metaphyseal, or distal articular)
* Age ≥18 years
* Indicated for definitive operative management at a single Level 1 trauma center

Exclusion Criteria:

* Revision procedures
* Temporizing procedures (irrigation and debridement, external fixation)
* Regular narcotic use
* Psychiatric illness
* Dementia
* Neuromuscular deficit
* Allergy/intolerance to cocktail ingredients
* Clinical status that precludes verbal pain assessment (e.g. major intracranial trauma)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Willey, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Busch CA, Whitehouse MR, Shore BJ, MacDonald SJ, McCalden RW, Bourne RB. The efficacy of periarticular multimodal drug infiltration in total hip arthroplasty. Clin Orthop Relat Res. 2010 Aug;468(8):2152-9. doi: 10.1007/s11999-009-1198-7. Epub 2009 Dec 18. PMID 20020333
- [Background] Kang H, Ha YC, Kim JY, Woo YC, Lee JS, Jang EC. Effectiveness of multimodal pain management after bipolar hemiarthroplasty for hip fracture: a randomized, controlled study. J Bone Joint Surg Am. 2013 Feb 20;95(4):291-6. doi: 10.2106/JBJS.K.01708. PMID 23302898

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peri-incisional Injection | Control (no Injection)
Started | 47 | 55
Completed | 45 | 50
Not Completed | 2 | 5
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peri-incisional Injection | Control (no Injection) | Total
Number analyzed (Participants) | 47 | 55 | 102
Age, Categorical [Count of Participants; unit: Participants] — Population: Although 102 subjects were randomized into the study, seven patients (2 in the injection group and 5 in the control group) were excluded following randomization because of early postoperative mortality (n = 1) and postoperative delirium (n = 6).
  Participants
    number analyzed (Participants) | 45 | 50 | 95
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 8 | 15 | 23
    >=65 years | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Although 102 subjects were randomized into the study, seven patients (2 in the injection group and 5 in the control group) were excluded following randomization because of early postoperative mortality (n = 1) and postoperative delirium (n = 6).
  years
    number analyzed (Participants) | 45 | 50 | 95
    (all) | 72.8 (15.2) | 70.0 (15.2) | 71.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Although 102 subjects were randomized into the study, seven patients (2 in the injection group and 5 in the control group) were excluded following randomization because of early postoperative mortality (n = 1) and postoperative delirium (n = 6).
  Participants
    number analyzed (Participants) | 45 | 50 | 95
    Female | 29 | 36 | 65
    Male | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United States | 47 | 55 | 102

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Assessment
Description: Patients will describe their current level of comfort on a 10 point scale while at rest. Zero corresponds to "no pain" and ten corresponds to "the most extreme possible pain." Visual analog scores will be collected by nursing staff who are blinded to the treatment allocation.
Time Frame: Pain assessment will be collected immediately prior to surgery (pre-op), immediately following surgery in the post-anesthesia care unit (PACU), and every 4 hours following surgery for the first two post-operative days (48 hours total; 4H-48H)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Peri-incisional Injection | Control (no Injection)
Number analyzed (Participants) | 45 | 50
units on a scale
  Pre-op | 5.0 [3.0 to 7.0] | 5.0 [2.0 to 7.0]
  PACU | 1.6 [0 to 4.0] | 3.2 [1.3 to 5.7]
  4H | 1.0 [0 to 3.0] | 5.0 [2.0 to 7.0]
  8H | 2.0 [0 to 4.0] | 5.0 [2.0 to 6.8]
  12H | 3.5 [0 to 5.0] | 5.0 [2.0 to 8.0]
  16H | 3.5 [2.0 to 5.8] | 4.0 [2.8 to 6.0]
  20H | 4.0 [2.0 to 6.0] | 4.0 [2.0 to 5.8]
  24H | 3.0 [2.0 to 5.8] | 4.0 [3.0 to 6.0]
  28H | 3.0 [0.8 to 5.0] | 3.5 [2.0 to 5.0]
  32H | 3.0 [1.0 to 4.0] | 5.0 [3.0 to 6.0]
  36H | 4.0 [1.0 to 5.0] | 4.0 [2.0 to 5.0]
  40H | 3.0 [2.0 to 5.0] | 3.5 [2.0 to 5.0]
  44H | 3.0 [0 to 5.0] | 4.0 [2.0 to 5.0]
  48H | 3.0 [1.0 to 5.0] | 3.0 [2.0 to 4.8]

2. Secondary Outcome: Total Narcotic Consumption
Description: Parenteral and oral narcotic agents will be utilized by patients for post-operative pain control per the standard of care. No alterations in narcotic prescription behavior will be observed for this study.
Time Frame: Narcotic consumption will be recorded every 8 hours for the first two post-operative days.
Measure: Mean (Inter-Quartile Range); unit: mg of morphine
Arm/Group | Peri-incisional Injection | Control (no Injection)
Number analyzed (Participants) | 45 | 50
mg of morphine | 5.0 [1.3 to 8.0] | 9.7 [3.9 to 15.6]

3. Other Pre Specified Outcome: Number of Participants With Medication-related Side Effects
Description: Patients will be monitored every 15 minutes in the recovery room and every 4 hours for the first two post-operative days by nursing personnel for medication side effects related to ropivacaine toxicity including blurred vision, hearing problems, transient peripheral paralysis, dizziness, convulsion, uncontrolled muscle contraction, hypotension, bradycardia, and new onset arrhythmia.
Time Frame: 48 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Peri-incisional Injection | Control (no Injection)
Number analyzed (Participants) | 45 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients will be monitored every 15 minutes in the recovery room and every 4 hours for the first two post-operative days by nursing personnel for Serious Adverse Events (SAE) and Other (Non Including Serious) Adverse Events (AEs).
Groups:
- Peri-incisional Injection: A 100 cc multimodal analgesic cocktail will be injected into the superficial and deep peri-incisional tissues after the completion of femur fracture fixation/instrumentation while the patient remains under general anesthesia and prior to wound closure. The cocktail includes 400 mg of 0.75% ropivacaine (53.33 mL), 0.6 mg of 1 mg/mL epinephrine (0.6 mL), 5 mg of 0.5 mg/mL morphine sulfate (10 mL), and 36.07 mL 0.9% sodium chloride solution. All infiltrations will be completed with a blunt trochar to minimize the risk of intravascular injection.
Arm/Group | Peri-incisional Injection | Control (no Injection)
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/55
Other Adverse Events (participants affected / at risk) | 0/47 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes